CLINICAL TRIAL: NCT07042269
Title: Comparative Effects of Respiratory Muscle Training Versus Aerobic Exercise on Cardiopulmonary Function in Older Adults: Determination of Temporal Adaptation Thresholds
Brief Title: Exploring the Time Effect of Respiratory Muscle Training on the Pulmonary Function of Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021096H
Record Dates: First submitted 2025-06-25; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Muscle Training; Aerobic Exercise; Older Adults; Cardiopulmonary Function
Keywords: Aerobic Exercise; Respiratory Muscle Training; Cardiopulmonary Function; Older Adults
MeSH Terms: interventions — Exercise; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): * Performed daily 10,000-step walking (5 days/week)
  * Exercise adherence was assessed using the Exercise Adherence Questionnaire
  Interventions: Behavioral: Aerobic Exercise
- Respiratory Muscle Training (RMT) Group (Experimental): * Performed 12-week progressive resistance training using the Lung Fitness breathing trainer (initial/moderate/high resistance levels)
  * Training protocol: 10 breaths/set, 3 sets/session (morning and evening), 5 days/week
  * Technique specification:
    1. Diaphragmatic breathing pattern
    2. Complete breath cycle = 1 repetition (inhalation ≤3s, exhalation ≤6s)
  * Resistance progression:
  * Initial level: Expiratory resistance - Level 1; Inspiratory resistance - Level 2
  * Moderate level: Expiratory resistance - Level 2; Inspiratory resistance - Level 3
  * High level: Expiratory resistance - Level 3; Inspiratory resistance - Level 4
  Interventions: Behavioral: Respiratory Muscle Training

INTERVENTIONS:
Behavioral: Aerobic Exercise — Performed daily 10,000-step walking (5 days/week)
  Arms: Aerobic Exercise Group
Behavioral: Respiratory Muscle Training — Performed 12-week progressive resistance training using the Lung Fitness® breathing trainer (initial/moderate/high resistance levels)
  Arms: Respiratory Muscle Training (RMT) Group

SUMMARY:
The goal of this clinical trial is to determine the effects of a 12-week respiratory muscle training (RMT) intervention on cardiopulmonary function and compare its efficacy with aerobic exercise in older adults. The main questions it aims to answer are:

* What are the effects of RMT compared to aerobic exercise on cardiopulmonary function?
* What is the minimal effective duration (temporal threshold) for observable physiological adaptations to RMT?
* To what extent are the training effects retained at 4-weeks post-intervention? Participants were randomly divided into RMT group and aerobic exercise group. The RMT group performed 12 weeks of progressive resistance training (initial, moderate, and high levels) using the Lung Fitness® breathing trainer, consisting of 10 breaths per set, 3 sets per session, twice daily (morning and evening), 5 days per week. The Aerobic Exercise group performed daily 10,000-step walking sessions 5 days per week, with exercise adherence assessed using the Exercise Adherence Questionnaire.

DETAILED DESCRIPTION:
30 subjects were finally included through the screening criteria. The names of all subjects were entered into Microsoft Excel 2016 and the RAND function was used to generate a random number between 0 and 1 for each subject, each random number being different. Subjects with an odd number of random numbers were assigned to the respiratory muscle training (RMT) group and those with an even number of random numbers were assigned to the aerobic exercise group. The final two intervention groups of 30 participants, were assigned and baseline testing was performed. Testing was repeated at five standardized time points (baseline, week 4, week 8, week 12 [post-intervention], and week 16 [post-detraining]).

The technical route of this study was to collect basic information about the study subjects, including age, height, weight, and to test the inspiratory muscle function, pulmonary function and the 6MWT of the study subjects. The RMT group performed 12 weeks of progressive resistance training (initial, moderate, and high levels) using the Lung Fitness® breathing trainer, consisting of 10 breaths per set, 3 sets per session, twice daily (morning and evening), 5 days per week. The aerobic exercise group performed daily 10,000-step walking sessions 5 days per week, with exercise adherence assessed using the Exercise Adherence Questionnaire.

Basic information and experimental data entry and organization were performed using Microsoft Excel 2016, and the results of all indicators measured before and after the experiment were analyzed and calculated in International Business Machines (IBM) SPSS Statistics 26.0. The data were tested for normality using the Shapiro-Wilk Test (Shapiro-Wilk Test). For the series conforming to the normal distribution, expressed as mean (Mean) and standard deviation (SD). Variables derived from inspiratory muscle function tests, pulmonary function tests, and 6MWT were analyzed for intergroup differences using paired-samples t-tests. Within-group comparisons across different time points in the RMT group were assessed via one-way repeated-measures analysis of variance (ANOVA) with Bonferroni post hoc correction. RPB and RPE were analyzed using nonparametric tests (Wilcoxon signed-rank test). Statistical significance was set at p < .05 (two-tailed). All data were tested for normality using the Shapiro-Wilk test prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60-75 years; Regardless of sex; Individuals classified as either physically inactive or habitual exercisers;

Exclusion Criteria:

* Individuals with cardiorespiratory diseases, hypertension, metabolic disorders, or other underlying medical conditions; Persons with impaired mobility, exercise contraindications, or inability to complete the exercise protocol; Inability to independently complete a Six-Minute Walk Test (6MWT) distance.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle function | Each subject was tested at five standardized time points (baseline, week 4, week 8, week 12 [post-intervention], and week 16 [post-detraining]).
  Inspiratory muscle function was quantified using a calibrated POWERbreathe K5 device (POWERbreathe International, Ltd., Southam, UK). Following standardized procedures [18], MIP and peak inspiratory flow (PIF) were recorded. Three technically acceptable maneuvers were performed at each session, with the highest value retained for analysis (coefficient of variation <10%).

SECONDARY OUTCOMES:
Pulmonary function | Each subject was tested at five standardized time points (baseline, week 4, week 8, week 12 [post-intervention], and week 16 [post-detraining]).
  Pulmonary function was conducted with a CHEST-H101 system (Chest M.I., Inc., Tokyo, Japan) calibrated daily, according to American Thoracic Society/European Respiratory Society (ATS/ERS) technical standards [19]. Parameters included VC, FVC, expiratory volume in one second (FEV1), and maximum expiratory flow rate (PEF). The best of three reproducible trials (within 150 mL or 5% variability) was selected.

OTHER OUTCOMES:
6MWT | Each subject was tested at five standardized time points (baseline, week 4, week 8, week 12 [post-intervention], and week 16 [post-detraining]).
  The 6MWT was administered on a 30 m indoor walkway with environmental controls (temperature 22 ± 1°C, humidity 50 ± 5%). Participants were instructed to "walk as far as possible" following ATS guidelines [20]. Standardized encouragement ("You're doing well, keep going") was provided during the final minute. The total distance walked was recorded to the nearest 0.5 m using a wheel-mounted measuring device. Immediately post-6MWT, dyspnea and leg fatigue were assessed using the modified Borg CR-10 scale: respiratory perceived exertion (RPE) and peripheral perceived exertion (PPE). Heart rate was continuously monitored via the Suunto Smart Sensor (Suunto Oy, Finland) chest strap, with HRmax defined as the highest 5 s average.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Xue Li, Doctor, Study Chair — Beijing Sports University; Xu Guo, Master, Principal Investigator — Beijing Sports University
Locations (1):
- Beijing Sports University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodrigues GD, Dal Lago P, da Silva Soares PP. Time-dependent effects of inspiratory muscle training and detraining on cardiac autonomic control in older women. Exp Gerontol. 2021 Jul 15;150:111357. doi: 10.1016/j.exger.2021.111357. Epub 2021 Apr 14. PMID 33864832